CLINICAL TRIAL: NCT04993378
Title: A Clinical Study Initiated by Investigator:Prospectively Predict the Efficacy of Precise Treatment of Gastrointestinal Tumors Based on Peripheral Blood Multi-omics Liquid Biopsy
Brief Title: Prospectively Predict the Efficacy of Treatment of Gastrointestinal Tumors Based on Peripheral Multi-omics Liquid Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Lin (Other)
Responsible Party: Sponsor-Investigator, Shen Lin, Director of GI oncology Affiliation: Peking University, Peking University
Organization: Peking University (Other)
Other Study IDs: CGOG-EV-1001
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Advanced Gastric Adenocarcinoma; Immunotherapy
Keywords: plasma-based liquid biopsy protein biomarker; extracellular vesicles; protein biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GC patients receiving immunotherapy
  Interventions: Device: EV-array

INTERVENTIONS:
Device: EV-array — Collect peripheral blood sample of 40 gastric cancer patients pre-treatment. Blood samples will be transferred to central lab to detect EV-score by EV-array. Tumor response evaluation will be performed after two cycles of chemotherapy by CT/MRI based on RECIST.
  Clinical data, including tumor stage, metastastic organ, regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
To vertify the function of EV-score on predicting & monitoring immunotherapeutic outcomes of GC

DETAILED DESCRIPTION:
Our previous work identified four plasma EV-derived proteins and combined them to generate a signature score that robustly predicting immunotherapeutic outcomes at baseline and dynamically monitoring disease progressions along with the whole treatment.

Hence in this stuty, we plan to recruit a prospective cohort to support our conclusions, and provide possible method to realize predicting and monitoring immunotherapeutic outcomes of GC.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Measurable disease according to the RECIST criteria
* Life expectancy of ≥3 month
* No prior chemotherapy of the study more than 4 weeks
* Immunotherapy regimens were included in the treatment

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study were enrolled by the Department of gastrointestinal oncology, Peking University Cancer Hospital & Institute for conventional therapy or clinical trials
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
EV-Score | EV-Score was detected, analysis and reported at the baseline of the treatment.
  EV-Score was calculated by the expression level of four tumor-associated proteins on plasma EV

SECONDARY OUTCOMES:
Survival significance of EV-Score | up to 3 years
  Analysis patients' survival with different EV-Score.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided